CLINICAL TRIAL: NCT05356598
Title: Impact of Peer-delivered Versus Authority-delivered Information on Help-seeking Intentions of ROTC Trainees
Brief Title: Help-seeking Intentions of ROTC Trainees
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UNLV-2022-55
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Help-Seeking Behavior; Musculoskeletal Injury
MeSH Terms: conditions — Help-Seeking Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peer-delivered (Experimental): The arm will receive an intervention in the form of a peer-delivered video promoting help-seeking for musculoskeletal injuries while in ROTC. This video will be presented by a current ROTC cadet.
  Interventions: Other: Peer-delivered Health Promotion Video
- Authority-delivered (Experimental): The arm will receive an intervention in the form of an authority-delivered video promoting help-seeking for musculoskeletal injuries while in ROTC. This video will be presented by a US Army Lieutenant Colonel who is currently a professor of military science for an ROTC battalion.
  Interventions: Other: Authority-delivered Health promotion video
- Control (Other): The arm will receive no true intervention. Participants in the control arm will watch a video of a US Army First Lieutenant exercising with no reference to musculoskeletal injuries or help-seeking behavior.
  Interventions: Other: Control Group Video

INTERVENTIONS:
Other: Authority-delivered Health promotion video — A video delivered by a US Army Lieutenant Colonel (authority figure) encouraging participants to seek help for musculoskeletal injuries experienced while in ROTC.
  Arms: Authority-delivered
Other: Peer-delivered Health Promotion Video — A video delivered by a US Army ROTC cadet (peer) encouraging participants to seek help for musculoskeletal injuries experienced while in ROTC.
  Arms: Peer-delivered
Other: Control Group Video — Video of a US Army First Lieutenant squatting, bench pressing, and deadlifting with voiceover. No mention of musculoskeletal injuries or help-seeking behavior.
  Other Names: Control
  Arms: Control

SUMMARY:
Online survey measuring pre-post stigma and intentions to seek care for musculoskeletal injuries using peer and authority-delivered health promotion videos.

DETAILED DESCRIPTION:
The survey will be hosted via QualtricsXM and accessible via an anonymous link. When participants open the survey, they will be presented with the survey's information sheet explaining the study's purpose and procedures. The information sheet will make it clear that completing the survey is voluntary and cadets may cease the survey at any time. Data from unfinished surveys will not be included in final analyses for any reports produced from this survey. Participants will complete demographics questions. Then, participants will answer injury reporting intentions and stigma questions, presented in a randomized order to reduce respondent fatigue. Participants will then watch a health promotion video that encourages reporting musculoskeletal injuries while in ROTC. Participants have the potential to be shown one of three videos: an officer-delivered health promotion, cadet-delivered health promotion, and a video of an officer exercising. Participants will be randomly assigned to one of the three videos using the in-built randomization function within Qualtrics. After watching the video, participants will answer the stigma and intentions questions again. After, participants will be asked to provide an email address that will be used to send them a link to complete the survey a second time. The follow-up portion will ask for their unique identifier as described above and have the participants answer the stigma and intentions questions again. All data will be de-identified when exporting responses from Qualtrics. No reference will be made to any individual participant in any way when presenting or reporting these data.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-39
* Actively participating in a college or university senior ROTC program (Army, Air Force, or Naval)

Exclusion Criteria:

* Anyone who does not meet inclusion criteria

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Stigma and Help-seeking Intentions Measured Before and After Health Promotion with Three-week Follow-up | Three weeks (baseline, immediately post intervention, and three weeks post intervention)
  Outcome will measure stigma and help-seeking intentions related to musculoskeletal injuries using an online survey. Survey items use a seven-point Likert scale where the most positive response is assigned the lowest number (1) while the most negative response is assigned the highest number (7).

CONTACTS AND LOCATIONS:
Overall Officials: Kara Radzak, PhD, Principal Investigator — University of Nevada, Las Vegas

IPD SHARING:
Plan to Share IPD: Undecided